CLINICAL TRIAL: NCT04421300
Title: Clinical Efficacy of Smile Exercise Versus 0.1% Hyaluronic Acid Sodium Eye Drops for Dry Eye Symptoms in Patients With Dry Eye Disease: a Randomized, Controlled, Non-inferiority Trial
Brief Title: A Randomized Study of Smile Exercise for Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020KYPJ010
Record Dates: First submitted 2020-06-01; First posted 2020-06-09 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Dry Eye; Keratoconjunctivitis Sicca; Eye Diseases; Corneal Diseases; Conjunctival Diseases
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca; Eye Diseases; Corneal Diseases; Conjunctival Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smile exercise (Experimental): smile exercise, 4 times a day，8 weeks
  Interventions: Behavioral: smile exercise
- 0.1% Sodium Hyaluronate Eye Drops (Active Comparator): 0.1% sodium hyaluronate, 4 times a day, 8 weeks.
  Interventions: Drug: 0.1% sodium hyaluronate eye drop

INTERVENTIONS:
Behavioral: smile exercise — Launch the "smile face recognition" APP on smart phone, after user guidance and pretest, a smile exercise will display on the phone, while facing the front camera on the phone, participant will do an exercise emphasizing facial movements, as exaggerated as possible. The exercise last for 8 weeks and 4 times a day
  Arms: smile exercise
Drug: 0.1% sodium hyaluronate eye drop — 0.1% sodium hyaluronate, 4 times a day, the time is in the morning, lunchtime, afternoon and evening. the interval between two training time is 2 hours, 1 hour before and after can be added or subtracted by users, 8 weeks.
  Arms: 0.1% Sodium Hyaluronate Eye Drops

SUMMARY:
The objective of the study is to evaluate the effectiveness of laughter therapy in relieving the symptoms of dry eye disease.

DETAILED DESCRIPTION:
The study is designed to: Test the hypothesis that smile exercise is an effective treatment for Dry Eye Disease (DED) . Better understand the status of emotion, quality of sleep and life in DED patient by describing and evaluating a comprehensive set of features and treatment over 2 months of observation in a well-characterized group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent approved by the Ethics Committee,
2. 18 to 45 years of age,
3. Meetting the dry eye diagnostic criteria of DEWs Ⅱ and demonstrating the following 2 condition in the same eye at screening and baseline visits (Same signs must present at both in Screening visit and Baseline visit). The same signs must be present in the same eye on both visits. The following parameters:.

   * Ocular Surface Disease Index (OSDI) score: 18-80 at and baseline visit.
   * Tear film break up time (TFBUT)<8s.
4. Best corrected visual acuity ≥10/20 in each eye
5. Intraocular pressure (IOP) ≥5mmHg and≤21mmHg in each eye
6. Women of child-bearing potential must agree to use a reliable method of contraception during study participation and must demonstrate a negative urine pregnancy test at the Screening Visit.
7. Feasible for all visits and willing to follow instructions from the study investigator.

Exclusion Criteria:

1. Corneal fluorescein staining present >5 score.
2. Contact lens wearing history:

   * Used contact lenses within last 14 days prior to the Screening Visit.
   * Unwilling to avoid using contact lenses druing the study.
3. Any corneal surgery within 12 months before Screening Visit .
4. Participation in other medical studies 3 months before screening Visit.
5. Current or previous diagnosis of any following ocular conditions in 3 months:

   i). acute allergic conjunctivitis ii). infection (e.g. bacterial, viral, protozoan or fungal infection of the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids) iii). inflammation (e.g., retinitis, macular inflammation, choroiditis, uveitis, scleritis, episcleritis, keratitis)
6. Eyelid abnormalities that affect lid function (e.g. lagophthalmos, blepharospasm, ectropion, entropion, severe trichiasis, etc.)
7. Extensive ocular surface scarring or condition that may compromise ocular surface integrity such as Stevens-Johnson syndrome, prior chemical burn, recurrent corneal erosions, persistent corneal epithelial defects, prior ocular trauma, etc.)
8. Currently diagnosis of glaucoma and under glaucoma medication or surgery treatment
9. Currently using, or intent to have any specific treatments for dry eye disease
10. Fluorescein sodium allergy
11. Pregnant, nursing, or lactating
12. Neurological or psychiatric disorders (moderate anxiety, depression and sleep disorders)
13. Uncontrolled ocular or systemic diseases
14. History of epilepsy .
15. The researchers did not consider the patient is appropriate for inclusion in this study
16. Cognitive or psychiatric defect that precludes informed consent or ability to perform requirements in the investigation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 299 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Change of Ocular Surface Disease Index (OSDI) Score | 12 weeks
  OSDI scores from 1, 2, 4, 6, 8, 10 and 12 weeks minus values from baseline. OSDI scores range from 0 to 100, score 0 indicating no ocular discomfort and higher scores indicating greater symptom severity. The minimal clinically significant change is 10 points.

SECONDARY OUTCOMES:
Proportion of Participants with 10 Points or More Decreased in OSDI | 12 weeks
  Proportion of participants with at least 10 points decreased from baseline in Ocular Surface Disease Index (OSDI).
Change from Baseline in Lipid layer thickness (LLT) | 12 weeks
  LLT from 1, 2, 4, 6, 8, 10 and 12 weeks minus values from baseline among eyes that qualified for the study. The interferometer LLT measurement is a non-invasively and objectively method that produces numeric value. The range of the value is 0-100+; lower value indicates thinner lipid layer.
Change in Non-invasive Tear film breakup time (NI-BUT) | 12 weeks
  In this measurement, NI-BUT is measured using the keratography machine. NI-BUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film. Change is record as the values at 1, 2, 4, 6, 8, 10 and 12 weeks minus values at baseline visit. Possible range of score is 0->20. Lower values indicate greater severity.
Change in Tear Meniscus Height (TMH) by Keratography | 12 weeks
  Assessment of the tear film meniscus is a quantitative measurement of tear film quantity. In this measurement, TMH is measured using the keratography machine. Change is the values at 1, 2, 4, 6, 8, 10 and 12 weeks minus values at baseline visit.
Change in Corneal Fluorescein Staining Score | 12 weeks
  Corneal Flourescein Staining Score from 1, 2, 4, 6, 8, 10 and 12 weeks minus values from baseline visit among eyes that quality that qualified for the study. Possible range of scores is 0-15; higher scores indicate more severe.
Change in Self-Rating Anxiety Scale (SAS) | 12 weeks
  Medical Outcomes from study 20-Item Self-Rating Anxiety Scale. This scale range is 0-100 with lower scores indicating better self-reported mental health. Change is the score at 4, 8 and 12 weeks minus the score at baseline visit.
Change in Self-Rating Depression Scale (SDS) | 12 weeks
  Medical Outcomes from study 20--Item Self-Rating Depression Scale. This scale range is 0-100 with lower scores indicating better self-reported mental health. Change is the score at 4, 8 and 12 weeks minus the score at baseline visit.
Change in Subjective Happiness Scale | 12 weeks
  A 4-item scale designed to measure subjective happiness. Each of item is completed by choosing one of 7 options that finish a given sentence fragment. Change is the score at 4, 8 and 12 weeks minus the score at baseline visit.
Change in Pittsburgh Sleep Quality Index (PSQI) | 12 weeks
  Change is the score at 4, 8 and 12 weeks minus the score at the baseline visits. Scores for each question range from 0 to 3, and the total PSQI scores range from 0 to 100.
Change in SF-36 Physical Health Subscale | 12 weeks
  Medical Outcomes from study 36-Item Short Form Health Survey (SF-36) Physical Health Subscale. Subscale range is 0-100, with higher scores indicating better self-reported physical health-related quality of life. Change is the score at 4, 8 and 12 weeks minus the score at baseline visit.
Change in SF-36 Mental Health Subscale | 12 weeks
  Medical Outcomes from study 36-Item Short Form Health Survey (SF-36) Mental Health Subscale. Change is the score at 4, 8 and 12 weeks minus the score at baseline visit.

OTHER OUTCOMES:
Change in Tear Cytokine Level | 12 weeks
  Change in levels of tear cytokines (mainly in inflammation cytokines, such as iL-17, TNF-alpha, etc.,). Change is the values from 8 and 12 weeks minus the the score at baseline visit.
Change in Lid Margin Abnormalities | 12 weeks
  Lid margin abnormalities were scored from 0 to 4 Change in lid margin abnormalities is the score from 4, 8 and 12 weeks minus the score at baseline visit.
Change in Meibum Quality | 12 weeks
  To evaluate meibum quality,five glands of the central part of the upper lid were assessed on a scale of 0-3 for each gland (total score range, 0-15).Change is the total score from 4, 8 and 12 weeks minus the score at baseline visit.
Change in Meibomian Gland Expressibility | 12 weeks
  The score of meibomian gland expressibility is range from 0-3. Change is the total score from 4, 8 and 12 weeks minus the score at baseline visit.
Change in Tear Film Break up Time, in Seconds (fluorescein staining) | 12 weeks
  Tear film break up time from1, 2, 4, 6, 8, 10 and 12 weeks minus values from baseline visit.
Change in Meibomian gland structure by Keratography | 12 weeks
  Change in Meibomian gland structure measured using the keratography machine. Change is the score from 8 and 12 weeks minus the values at baseline visit

CONTACTS AND LOCATIONS:
Locations (1):
- Zhonshan Ophthalmic Centre, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Liao Y, Zhang SY, Jin L, Congdon N, Fan Z, Zeng Y, Zheng Y, Liu Z, Liu Y, Liang L. Effect of laughter exercise versus 0.1% sodium hyaluronic acid on ocular surface discomfort in dry eye disease: non-inferiority randomised controlled trial. BMJ. 2024 Sep 11;386:e080474. doi: 10.1136/bmj-2024-080474. PMID 39260878